CLINICAL TRIAL: NCT03874897
Title: An Open Label, Single/Multiple Dose Exploratory Clinical Study to Evaluate the Safety, Efficacy, and Cytokinetics of Autologous Humanized Anti-claudin18.2 Chimeric Antigen Receptor T Cell in Advanced Solid Tumor Subjects
Brief Title: Chimeric Antigen Receptor T Cells Targeting claudin18.2 in Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT041-CG4006
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced solid tumor; claudin18.2; CAR-T cell therapy
MeSH Terms: interventions — spartalizumab; toripalimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CAR-CLDN18.2 T-Cells (Experimental): The subjects enrolled will be sequentially assigned to the corresponding dose level.
  Interventions: Drug: CAR-CLDN18.2 T-Cells
- Cohort 1 (Experimental): CT041 monotherapy in patients with GI cancers who failed standard chemotherapy
  Interventions: Drug: CAR-CLDN18.2 T-Cells
- Cohort 2 (Experimental): CT041 plus anti-PD1 therapy in patients with GI cancers who failed standard chemotherapy
  Interventions: Drug: CAR-CLDN18.2 T-Cells; Drug: PD-1 Monoclonal Antibody
- Cohort 3 (Experimental): CT041 sequential treatment after first-line therapy in GC/GEJ
  Interventions: Drug: CAR-CLDN18.2 T-Cells; Drug: Chemotherapy
- Cohort 4 (Experimental): prior treatment failure to anti-CLDN18.2 monoclonal antibody
  Interventions: Drug: CAR-CLDN18.2 T-Cells

INTERVENTIONS:
Drug: CAR-CLDN18.2 T-Cells — Preconditioning with fludarabine, cyclophosphamide, based chemotherapy regimen at sub-clinical doses
  • Chimeric Antigen Receptor T Cells Targeting Claudin18.2
  Other Names: Chimeric Antigen Receptor T Cells Targeting Claudin18.2
Drug: PD-1 Monoclonal Antibody — Chimeric Antigen Receptor T Cells Targeting Claudin18.2 with PD-1
  Other Names: Toripalimab
  Arms: Cohort 2
Drug: Chemotherapy — First-line systemic therapy according to physician's choice
  Arms: Cohort 3

SUMMARY:
An open label, single/multiple dose exploratory clinical study to evaluate the safety, efficacy, and pharmacokinetics of autologous humanized anti-claudin18.2 chimeric antigen receptor T cell in advanced solid tumor.

DETAILED DESCRIPTION:
This study is an open, single/multiple infusion, dose escalation/dose regimen finding study to assess the safety and pharmacokinetics of CAR-CLDN18.2 T cell therapy, and to obtain the preliminary efficacy results in subjects who have been diagnosed with advanced solid tumor with positive claudin 18.2 expression and failed to standard systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, male or female;
2. Subjects with pathologically confirmed solid tumors (ie, advanced gastric cancer, esophagogastricgastroesophageal junction cancer, and pancreatic cancer) and have been failed to at least first-one prior line of systemic treatment;
3. Tumor tissue samplessample was positive for claudin 18.2 positive through for claudin18.2 IHC staining;assay(≥2+, and ≥40%);
4. Estimated life expectancy > 12 weeks;
5. According to the RECIST 1.1, there is at least one measurable or unmeasurable tumor lesionslesion；
6. ECOG physical status score 0 ~ 1, within 24 hours prior to apheresis, and at baseline (prior to pre-treatment);
7. Sufficient venous access for mononuclear cell collection (abbreviation: apheresis)
8. Subjects should have adequate organ functions before screening and pre-treatment (at baseline).
9. Female subjects of childbearing age must undergo a serum pregnancy test at screening and prior to preconditioning and the results must be negative, and are willing to use a very effective and reliable method of contraception within 1 year after the last study treatment. The methods that can be used are: bilateral tubal ligation / bilateral salpingectomy or bilateral tubal occlusion; or approved oral, injection or hormone-imparting contraceptive methods; or barrier contraceptive method: containing spermicidal foam / Gel/film/cream/suppository condom or occlusive cap (diaphragm or cervix/cap);
10. Men who have actively sexual intercourse with women with child-bearing potential, must agree to use barrier-based contraception if they have no vasectomy, for example, a condom containing a spermicidal foam/gel/film/paste/suppository, or use a contraceptive method for their spouse (see article 9 of the inclusion criteria). Moreover, all men are absolutely forbidden to donate sperm within 1 year after receiving the last study treatment infusion；
11. Subject participates in this clinical trial and sign Informed Consent Form voluntarily.

Exclusion Criteria:

1. Pregnant or lactating women;
2. HIV, Treponema pallidum or HCV serologically positive;
3. Any uncontrollable active infection, including but not limited to active tuberculosis, HBV infection (HBsAg positive, or HBcAb positive and HBV DNA positive);
4. Subjects have clinically significant thyroid dysfunction determined by investigator (serum thyroid hormone assays TT4, TT3, FT3, FT4, and serum thyroid stimulating hormone TSH) which is not suitable for entering into the study;
5. The side effects caused by the previous treatment of the subjects did not return to CTCAE ≤1; except hair loss and, hyperpigmentation or other tolerable events determined by investigator or laboratory abnormalities allowed by the protocol;
6. Subjects who are using steroidshave recieved ≥15 mg/day glucocorticoid systemically currently within 7 days prior to apheresis; those using inhaled steroids recently or currently are not excluded;
7. Previously allergic to immunotherapy and related drugs, history of severe allergiespreconditioning drug such as cyclophosphamide, fludarabine, or allergiestocilizumab or allergic to components of CT041CAR-CLDN18.2T injection, allergic to β-lactam antibiotics;the CT041 infusion;
8. Previously received any chimeric antigen receptor-modified T-cells(including CAR-T、TCR-T) .
9. Subjects have untreated or symptomatic brain metastases;
10. Subjects have central or extensivelywith centralcor diffused metastases in lung and .extensiveor diffused metastases in liver;liveror with rapid tumor progression since screening period evaluated by the investigator preconditioning (at baseline)；
11. The largest target tumor lesion>4cm
12. Subjects with unstable or active ulcers and gastrointestinal bleeding currently;
13. Subjects with a history of organ transplantation or awaiting organ transplantation;
14. Subjects requiring anticoagulant therapy;
15. Subjects requiring continuous anti-platelet therapy;
16. Subjects who have undergone major surgery or significant trauma within 4 weeks prior to apheresis, or who are expected to undergo major surgery during the study;
17. There are no other serious diseases that may limit subjects' participation in this trial;
18. The investigator assessed that the subject was unable or unwilling to comply with the requirements of the study protocol;
19. Blood oxygen saturation ≤ 95% before pre-treatmentapheresis or preconditioning (accept finger oxygen detection method);
20. Prior to pretreatmentpreconditioning, subjects developed, including but not limited to, new arrhythmias that could not be controlled with drugs, hypotension requiring pressor agent, bacterial, fungal or viral infections that required intravenous antibiotics. Creatinine clearance rate <40mL / min; The investigator judges that the subject is not suitable for continuing the trial. Subjects who use antibiotics to prevent infection can continue the trials if judged by the investigator;
21. The subject has a central nervous system disease sign or an abnormal neurological test result with clinical significance;
22. The subject is currently suffered from or have suffered from other incurable malignant tumors within previous 3 years, except in situ cervical cancer or skin basal cell cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days of single infusion
  Safety
Maximum tolerated dose (MTD) | 28 days of single infusion
  tolerability

SECONDARY OUTCOMES:
Pharmacokinetics (the number of cell copies and cell persistence duration in peripheral blood) | 26 weeks
  CAR-CLDN18.2 DNA in peripheral blood detected by q-PCR at each visit after infusion
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 1 year
  Adverse events occurring through 26 weeks and 12 months post infusion of CAR-CLDN18.2 T-Cell infusion, such as abnormalities or changes in laboratory examinations, physical examinations, vital signs, etc.
Antitumor efficacy-Progression-free survival (PFS) | 1 year
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-Duration of response (DOR) | 1 year
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause
Antitumor efficacy-Duration of disease control (DDC) | 1 year
  The period from the first evaluation of clinical benefit to the first evaluation of PD or any cause of death.
Antitumor efficacy-Overall survival (OS) | 1 years
  The period from the first infusion to any cause of death
Antitumor efficacy-Objective response rate (ORR) | 1 year
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR, the subjects should confirm it no less than 4 weeks after the first evaluation
Antitumor efficacy-Disease control rate (DCR) | 1 year
  The number of cases in which response are achieved from the start of cell infusion/the total number of evaluable cases (%).
Long term survival follow up | 15 years
  The period from the first infusion to any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Department of GI Oncology, Peking University Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital , Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Li J, Liu L, Tao M, Han Z, Ma M, Jiang L, Liu C, Liu D, Zhang P, Zhang M, Xue R, Gong J, Zhang X, Shen L, Qi C. Impact of concomitant medications on efficacy of CLDN18.2-specific CAR-T cell therapy in advanced gastric cancer. Br J Cancer. 2026 Feb;134(3):439-446. doi: 10.1038/s41416-025-03289-7. Epub 2025 Nov 29. PMID 41318814
- [Derived] Li J, Tao M, Liu L, Liu C, Ma M, Liu D, Zhang P, Zhang M, Xue R, Gong J, Zhang C, Zhang X, Shen L, Qi C. Peripheral blood neutrophils contribute to Claudin18.2-specific CAR-T cell treatment resistance in advanced gastric cancer. Br J Cancer. 2025 Jun;132(12):1167-1176. doi: 10.1038/s41416-025-03015-3. Epub 2025 Apr 17. PMID 40246985
- [Derived] Qi C, Liu C, Gong J, Liu D, Wang X, Zhang P, Qin Y, Ge S, Zhang M, Peng Z, Zhou J, Lu Z, Lu M, Cao Y, Yuan J, Wang Y, Wang Z, Xue R, Peng X, Wang Y, Yuan D, Li J, Zhang X, Shen L. Claudin18.2-specific CAR T cells in gastrointestinal cancers: phase 1 trial final results. Nat Med. 2024 Aug;30(8):2224-2234. doi: 10.1038/s41591-024-03037-z. Epub 2024 Jun 3. PMID 38830992
- [Derived] Qi C, Zhang P, Liu C, Zhang J, Zhou J, Yuan J, Liu D, Zhang M, Gong J, Wang X, Li J, Zhang X, Li N, Peng X, Liu Z, Yuan D, Baffa R, Wang Y, Shen L. Safety and Efficacy of CT041 in Patients With Refractory Metastatic Pancreatic Cancer: A Pooled Analysis of Two Early-Phase Trials. J Clin Oncol. 2024 Jul 20;42(21):2565-2577. doi: 10.1200/JCO.23.02314. Epub 2024 May 24. PMID 38788174
- [Derived] Qi C, Xie T, Zhou J, Wang X, Gong J, Zhang X, Li J, Yuan J, Liu C, Shen L. CT041 CAR T cell therapy for Claudin18.2-positive metastatic pancreatic cancer. J Hematol Oncol. 2023 Sep 9;16(1):102. doi: 10.1186/s13045-023-01491-9. PMID 37689733
- [Derived] Qi C, Gong J, Li J, Liu D, Qin Y, Ge S, Zhang M, Peng Z, Zhou J, Cao Y, Zhang X, Lu Z, Lu M, Yuan J, Wang Z, Wang Y, Peng X, Gao H, Liu Z, Wang H, Yuan D, Xiao J, Ma H, Wang W, Li Z, Shen L. Claudin18.2-specific CAR T cells in gastrointestinal cancers: phase 1 trial interim results. Nat Med. 2022 Jun;28(6):1189-1198. doi: 10.1038/s41591-022-01800-8. Epub 2022 May 9. PMID 35534566